CLINICAL TRIAL: NCT03806452
Title: Multicentre Randomized Double-blind Placebo-controlled Study to Evaluate the Effect on Albuminuria of 6 Months Treatment With Hydroxycarbamide (Siklos®) or a Placebo in Adults With Sickle Cell Disease:
Brief Title: SIKAMIC (SIklos on Kidney Function and AlbuMInuria Clinical Trial)
Acronym: SIKAMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIK-FR-17-1
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: albuminuria; hydroxycarbamide
MeSH Terms: conditions — Anemia, Sickle Cell; Albuminuria | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxycarbamide (Experimental): Hydroxycarbamide will be supplied as 100 mg or 1000 mg film-coated tablets. The posology will be based on the patient's body weight (bw). Hydroxycarbamide will be prescribed at a dose of 15 mg/kg bw/day and will be adminitered for 6 months.
  Hydroxycarbamide will be administered for 12 months for patients qualified as responders willing to continue to participate in the trial.
  Interventions: Drug: Hydroxycarbamide
- Placebo (Placebo Comparator): Placebo will be supplied as 100 mg or 1000 mg film-coated tablets. The posology will be based on the patient's body weight (bw). Placebo will be prescribed at a dose of 15 mg/kg bw/day and will be adminitered for 6 months.
  Hydroxycarbamide will be administered for 12 months for patients qualified as responders willing to continue to participate in the trial.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Hydroxycarbamide — Hydroxycarbamide tablets of 100 and 1000 mg
  Other Names: Siklos
  Arms: Hydroxycarbamide
Drug: Placebo Oral Tablet — Placebo tablets of 100 and 1000 mg to mimic hydroxycarbamide tablets
  Arms: Placebo

SUMMARY:
The purpose of this phase IIb, international, multicentre, double-blind, randomised, placebo-controlled study is to determine the effect of hydroxycarbamide on albuminuria after 6 months of treatment in SCD adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (ICF) by a legally competent patient.
2. Patients above 18 years.
3. Patients with HbSS or HbSβ0 SCD.
4. Patients with a value of albuminuria, assessed by ACR, over 3 mg/mmol and inferior to 100 mg/mmol confirmed by 3 positive urine samples taken one day apart.
5. Female patients of childbearing potential or postmenopausal female with last period < 12 months before screening agreeing to use a highly effective form of contraception (oral, injected or implanted hormonal contraception, intrauterine device, diaphragm, condom) during the trial and for 3 months after hydroxycarbamide discontinuation.
6. Male patients with partners of childbearing potential agreeing to use a highly effective contraception during the trial and for 3 months after hydroxycarbamide discontinuation. Men with pregnant or lactating women should be advised to use a barrier method of contraception (condom) to prevent the foetus or breastfed infant from exposure to hydroxycarbamide.
7. Patients who are covered by insurance scheme according to local regulatory requierements.

Exclusion Criteria:

1. Patients who had severe VOC requiring hospitalisation or ACS within the last 4 weeks preceding screening visit.
2. Patients treated with hydroxycarbamide for any reason within the previous 6 months.
3. Patients who have had chronic blood transfusion or transfusion in the last 3 months.
4. Patients with a history of hypertension (systolic blood pressure ≥ 140 or diastolic blood pressure ≥ 90 mmHg) treated with antihypertensive agent belonging to pharmacological class of RAS inhibitor.
5. Patients who have symptoms suggestive of urinary tract infection or patients with gross haematuria.
6. Patients with a concomitant primary kidney disease.
7. Patients with any systemic condition that could result in a glomerulopathy not related to SCD (e.g. diabetes mellitus, active hepatitis B or C infections, HIV infection, systemic lupus erythematosus, inflammatory arthropathies).
8. Patient with a stage 3, 4 or 5 chronic kidney disease (eGFR < 60 mL/min per 1.73 m2).
9. Patients with eGFR ≥ 140 ml/min/1,73m² due to the lack of information regarding the magnitude, direction and significance of the trends in eGFR evolution that could be expected in this population
10. Patients requiring long-term treatment with drugs potentially nephrotoxic (see non-exhaustive list).
11. Patients requiring ACE inhibitors or ARBs within the 3 months before inclusion regardless of the indication.
12. Patients requiring long-term treatment with non-steroid anti-inflammatory drugs.
13. Patients who have a treatment which can modify the kidney function (see non-exhaustive list) in the last 3 months.
14. Patients known to be infected with HIV.
15. Female patients who are pregnant or lactating.
16. Unreliable patients including non-compliant patients, patients with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as patients unwilling to give informed consent or to abide by the requirements of the protocol.
17. Simultaneous participation in other clinical trials on an investigational medicinal product or previous participation within 30 days before inclusion.
18. Persons in detention by judicial or administrative decision.
19. Patients with chronic conditions that upon investigator judgment may lead to a limited life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Bartolucci, Pr, Principal Investigator — Henri Mondor University Hospital; Vincent Audard, Pr, Study Chair — Henri Mondor University Hospital
Locations (21):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire (CSRS), Abidjan, Côte d’Ivoire
- France (16):
  - CHU d'Angers, Angers
  - Hôpital Saint-André, Bordeaux
  - CHRU Brest, Brest
  - Hôpital Louis Mourier, Colombes
  - Pablo Bartolucci, Créteil
  - Hopital Edouard Herriot, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital européen Georges-Pompidou, Paris
  - Hôpital Saint-Antoine, Paris
  - Service de biothérapie, consultation hématologie-drépanocytose hôpital Necker, Paris
  - CHU la Miletrie, Poitiers
  - Hôpital Robert Debré CHU Reims, Reims
  - Hopital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - Centre Hospitalier Delafontaine, Saint-Denis
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- CHU Pointe-à-Pitre/Abymes, Pointe-à-Pitre, Guadeloupe
- Centre de Recherche et de Lutte contre la Drépanocytose de Bamako (CRLD), Bamako, Mali
- CHU Martinique, Le Lamentin, Martinique
- Service d'Hématologie Clinique, Centre National de Transfusion sanguine, Université Cheikh Anta Diop, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 28 May 2019 to 30 May 2024, 86 patients were included in the study in the mITT population and analysed in France and Africa (Mali, Ivory Coast and Senegal).
Groups:
- Hydroxycarbamide: Hydroxycarbamide will be supplied as 100 mg or 1000 mg film-coated tablets. The posology will be based on the patient's body weight (bw). Hydroxycarbamide will be prescribed at a dose of 15 mg/kg bw/day and will be adminitered for 6 months.
  Hydroxycarbamide will be administered for 12 months for patients qualified as responders willing to continue to participate in the trial.
  Hydroxycarbamide: Hydroxycarbamide tablets of 100 and 1000 mg
- Placebo: Placebo will be supplied as 100 mg or 1000 mg film-coated tablets. The posology will be based on the patient's body weight (bw). Placebo will be prescribed at a dose of 15 mg/kg bw/day and will be adminitered for 6 months.
  Hydroxycarbamide will be administered for 12 months for patients qualified as responders willing to continue to participate in the trial.
  Placebo Oral Tablet: Placebo tablets of 100 and 1000 mg to mimic hydroxycarbamide tablets
Period: Initial Treatment Period
Arm/Group | Hydroxycarbamide | Placebo
Started | 46 | 40
Completed | 44 | 38
Not Completed | 2 | 2
Period: Responders Extended Treatment Period
Arm/Group | Hydroxycarbamide | Placebo
Started | 18 | 15
Completed | 15 | 9
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxycarbamide | Placebo | Total
Number analyzed (Participants) | 46 | 40 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: one patient with missing information
  years
    number analyzed (Participants) | 45 | 40 | 85
    (all) | 30.3 (10.0) | 30.0 (8.7) | 30.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Continent of origin: Africa - America | 45 | 40 | 85
  Continent of origin: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Senegal | 17 | 12 | 29
  Mali | 12 | 8 | 20
  Guadeloupe | 0 | 1 | 1
  Côte D'Ivoire | 5 | 4 | 9
  Martinique | 1 | 0 | 1
  France | 11 | 15 | 26
SCD genotype [Count of Participants; unit: Participants]
  HbSS | 43 | 37 | 80
  HbSbeta0 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving at Least a 30% Decrease in ACR Baseline Value
Description: The primary endpoint of this study is the proportion of patients in the hydroxycarbamide and placebo groups achieving at least a 30% decrease in ACR baseline value at 6 months after treatment initiation. Patients who do not achieve at least a 30% decrease of the ACR baseline value at month 6 will be considered non-responders.
Time Frame: 6 months
Population: 3 patients in the hydroxycarbamide arm and 2 patients in the placebo arm do not have any measure at 6 months and so were not part of this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
Participants | 18 | 15

2. Secondary Outcome: Absolute Mean Changes in eGFR Value
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
ml/min/1.73m2 | 3.2 (18.5) | -1.0 (13.8)

3. Secondary Outcome: Absolute Mean Changes in ACR Value
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/mmol
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
mg/mmol | 3.5 (19.7) | 1.0 (13.1)

4. Secondary Outcome: Proportion of Patients With a Shift From Macroalbuminuria to Microalbuminuria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
Participants | 1 | 2

5. Secondary Outcome: Proportion of Patients With a Shift From Microalbuminuria to Normoalbuminuria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 8
Participants | 10 | 7

6. Secondary Outcome: Proportion of Patients With a Shift From Macroalbuminuria to Normoalbuminuria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
Participants | 1 | 0

7. Secondary Outcome: Proportion of Patients With a Shift From Microalbuminuria to Macroalbuminuria
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
Participants | 3 | 3

8. Secondary Outcome: Absolute Mean Changes of Systolic Blood Pressure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 40 | 34
mmHg | 2.8 (10.7) | 2.2 (13.1)

9. Secondary Outcome: Absolute Mean Changes of Body Weight
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 37
kg | 2.2 (3.0) | -0.3 (2.1)

10. Secondary Outcome: Absolute Mean Changes of Diastolic Blood Pressure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 40 | 35
mmHg | 2.5 (13.3) | -1.0 (12.9)

11. Secondary Outcome: Absolute Mean Changes of Heart Rate Measure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 41 | 37
beats/minute | -2.1 (11.3) | 2.4 (12.5)

12. Secondary Outcome: Absolute Mean Changes in White Blood Cells Count
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 37
cells/mm3 | -3659.6 (3524.4) | -228.4 (2982.1)

13. Secondary Outcome: Absolute Mean Changes in Platelets Count
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 37
10^9 platelets per liter | -49.3 (150.9) | -16.0 (83.5)

14. Secondary Outcome: Absolute Mean Changes in Mean Corpuscular Volume
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 37
fL | 15.1 (10.8) | -0.3 (3.4)

15. Secondary Outcome: Absolute Mean Changes in Mean Corpuscular Haemoglobin Concentration
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 33
g/L | 1.7 (15.8) | -4.8 (16.4)

16. Secondary Outcome: Absolute Mean Changes in Mean Corpuscular Haemoglobin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 34
pg | 5.5 (4.0) | -0.8 (1.6)

17. Secondary Outcome: Absolute Mean Changes in Hemoglobin Count
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 44 | 36
g/L | 12 (11.3) | -2.2 (6.1)

18. Secondary Outcome: Absolute Mean Changes in Foetal Hemoglobin Count
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 24 | 24
percentage of hemoglobin | 8.5 (8.8) | 0.3 (1.9)

19. Secondary Outcome: Absolute Mean Changes in Free Hemoglobin Count
Time Frame: 6 months and 12 months for responder patients willing to continue the study after month 6.
Reporting Status: Not Posted

20. Secondary Outcome: Absolute Mean Changes in Dense Red Blood Cells Percentage
Time Frame: 6 months and 12 months for responder patients willing to continue the study after month 6.
Reporting Status: Not Posted

21. Secondary Outcome: Absolute Mean Changes in Endogenous Erythropoietin Count
Time Frame: 6 months
Population: Very few patients have an evaluation of endogenous erythropoietin count. Only 3 in hydroxycarbamide group and 6 in placebo group
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 3 | 6
U/L | -8.2 (22.1) | 17.4 (37.1)

22. Secondary Outcome: Absolute Mean Changes in Ferritin Count
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 41 | 35
µg/L | 28.1 (664.2) | -8.0 (404.3)

23. Secondary Outcome: Absolute Mean Changes in Lactate Dehydrogenase
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 42 | 38
U/L | -170.5 (349.4) | -1.8 (220.9)

24. Secondary Outcome: Absolute Mean Changes in Aspartate Aminotransferase
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
U/L | -8.7 (19.2) | -1.0 (10.9)

25. Secondary Outcome: Absolute Mean Changes in Alanine Amino Transferase
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 43 | 38
U/L | -1.7 (51.2) | -0.2 (13.7)

26. Secondary Outcome: Absolute Mean Changes in Blood Urea Nitrogen
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 42 | 36
mmol/L | -0.5 (6.4) | 0.5 (2.6)

27. Secondary Outcome: Absolute Mean Changes in Conjugated Bilirubin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 39 | 35
µmol/L | -0.7 (33.8) | -1.9 (9.8)

28. Secondary Outcome: Absolute Mean Changes in Total Bilirubin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 40 | 35
µmol/L | -8.9 (106.5) | 4.7 (30.1)

29. Secondary Outcome: Absolute Mean Changes in Reticulocytes
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Hydroxycarbamide | Placebo
Number analyzed (Participants) | 40 | 36
cells/mm3 | -116082.5 (168548.6) | -35336.1 (108156.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Hydroxycarbamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 2/40
Serious Adverse Events (participants affected / at risk) | 5/46 | 7/40
Other Adverse Events (participants affected / at risk) | 30/46 | 29/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxycarbamide (N=46) | Placebo (N=40)
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
HEPATOBILIARY PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BONE INFARCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxycarbamide (N=46) | Placebo (N=40)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
ASTHENIA (General disorders) | 2 (2) | 5 (5)
CHEST PAIN (General disorders) | 1 (1) | 4 (5)
PYREXIA (General disorders) | 4 (6) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (6) | 3 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 3 (3)
HEADACHE (Nervous system disorders) | 8 (9) | 5 (6)
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
VERTIGO (Ear and labyrinth disorders) | 3 (3) | 5 (5)
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03806452/Prot_SAP_000.pdf